CLINICAL TRIAL: NCT05710029
Title: Cortical Processes During Walking Post-stroke
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB202202100
Record Dates: First submitted 2023-01-10; First posted 2023-02-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute; Walking, Difficulty
Keywords: Walking; Stroke; EEG; Assistance
MeSH Terms: conditions — Stroke; Mobility Limitation; Helping Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to use novel mobile imaging techniques with high-density electroencephalography (EEG) to quantify cortical processes synchronized to the biomechanics of walking. Here, the study has two aims - the primary aim is to quantify the cortical processes that contribute to gait dysfunction early post-stroke, and the second aim is to determine how cortical processes are mediated by mechanical assistance during early gait training post-stroke.

Participants will wear an electroencephalography (EEG) cap to measure brain activity and other non-invasive physiological sensors. Participants will be asked to perform different tasks, such as walking at different speeds and walking with different levels of body weight support.

DETAILED DESCRIPTION:
This study will recruit 15 subacute post-stroke individuals and 15 age-matched neurotypical individuals between the age of 18-80 years old.

ELIGIBILITY:
Inclusion Criteria for post-stroke patients:

* Participants will have a unilateral brain lesion within six months prior to participation in this project;
* Paresis confined to one side;
* Ability to walk for 10 meters continuously;
* Absence of severe cognitive dysfunction as demonstrated by a Mini-Mental score greater than 24;
* Absence of severe concurrent medical problems;
* Ability to provide informed consent.

Exclusion Criteria for age-matched adults:

* Any major neurological, cardiovascular, orthopedic, and psychiatric diagnoses

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Post-stroke participants (age 18-80), age-matched adults (age 18-80)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Brain activity during walking measured by EEG | through study study completion, an average of 2 years
  Changes in brain activity during walking with different levels of weight support
Brain activity during walking measured by EEG | through study study completion, an average of 2 years
  Differences in brain activity during walking between people post-stroke and neurotypical individuals

CONTACTS AND LOCATIONS:
Overall Officials: Chang Liu, PhD, Principal Investigator — University of Florida; Daniel Ferris, PhD, Principal Investigator — University of Florida; Dorian Rose, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Share deidentified data on an online repository